CLINICAL TRIAL: NCT06180746
Title: Study of the Conditions of the Effects of Health Mediation on Underserved Populations' Healthcare Utilization
Brief Title: Study of the Conditions of the Effects of Health Mediation on Underserved Population
Acronym: ECEMSo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2020/70
Record Dates: First submitted 2023-12-04; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Mediation
Keywords: Healthcare utilization; Health mediation; Cancer screening; Complex intervention; realist evaluation; study protocol; underserved populations
MeSH Terms: conditions — Negotiating

STUDY DESIGN:
Intervention Model Description: longitudinal mixed-method intervention study with a multi-center, multi-case explanatory sequential design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ECEMSo intervention (Experimental): This group is composed of health mediators, the people living in informal housing they support and stakeholders. The ECEMSo intervention will be implemented in this group
  Interventions: Behavioral: Knowledge mobilization to facilitate the structuring of health mediation
- Group 2 : No intervention (No Intervention): This group is composed of health mediators, the people living in informal housing they support and stakeholders. The ECEMSo intervention will not be implemented in this group.
- Group 3 : No intervention (No Intervention): This group is composed of health workers, social workers, the people living in informal housing they support and stakeholders. The ECEMSo intervention will be implemented in this group.

INTERVENTIONS:
Behavioral: Knowledge mobilization to facilitate the structuring of health mediation — The ECEMSo intervention involves knowledge mobilization to facilitate the structuring of health mediation throughout French territory, and the development of a co-designed effective action plan to facilitate cancer screening uptake by people living in informal housing.
  The action plan will, consider territorial specificities at the regional level. The ECEMSo project team will organize a seminar and three workshops. The aim of the seminar and workshops is to mobilize knowledge to facilitate i) the structuring of health mediation in the regions, and ii) the development of an action plan with health mediators and other stakeholders to foster organized cancer screenings uptake by underserved people. This action plan must match with the needs of people living in informal housing, and must be coordinated, suitable and feasible to implement, in terms of knowledge about people living in informal housing specificities and specific local collaborations
  Arms: ECEMSo intervention

SUMMARY:
The investigators are conducting a longitudinal mixed-method intervention study with a multi-center, multi-case explanatory sequential design. The ECEMSo study aims to identify the impact of health mediation on fostering healthcare utilization, in particular organized cancer screening uptake, by underserved populations living in informal housing in France.

DETAILED DESCRIPTION:
Health mediation may foster underserved populations' healthcare utilization. No study to date has demonstrated its effectiveness in an experimental context. The ECEMSo case study aims to identify the impact of health mediation on fostering healthcare utilization - in particular organized cancer screening uptake - by underserved populations living in informal housing in France.

Grounded in a theory-based framework, the ECEMSo case study is a longitudinal mixed-method intervention study with a multi-center, multi-case explanatory sequential design. The study population comprises various participant profiles including health mediators, health workers, social workers, people living in informal housing whom these professionals support, and other stakeholders concerned with underserved populations' health issues. Participants will be recruited in several French regions and divided into three mixed participant profile groups. In group 1, health mediation and the ECEMSo intervention will be implemented. This intervention comprises knowledge mobilization to facilitate the structuring of health mediation throughout France, and the development of an action plan to facilitate cancer screening uptake by people living in informal housing. In group 2, only health mediation will be implemented (i.e., no ECEMSo intervention). In group 3, neither health mediation nor the ECEMSo intervention will be implemented, but health and social workers will implement other health system navigation interventions.

Quantitative and qualitative data will be collected by interviewers through face-to-face questionnaires, interviews, observations, focus groups, and tracking tables of health mediation activities over six months. Data collection will be based on the health mediation conceptual framework.

ELIGIBILITY:
People living in informal housing

Inclusion criteria:

* Living on the streets, in a shanty house, squat or caravan
* Living in an area covered by one of care structures participating in the ECEMSo study
* Being over 18 years old
* Being able to understand the detailed information provided about the ECEMso study

Exclusion criteria:

* Suffering from cognitive and/or psychiatric disorders
* Being under guardianship or curatorship

Health mediators, heal workers, socials workers

Inclusion criteria:

* Being a health mediator, a health worker or a social worker belonging to one of the study's participation care structures
* Providing support to people living in informal housing

Exclusion criteria: No

Stakeholder:

Inclusion criteria: Being an actor concerned or involved with the issues and needs of people living in informal housing

Exclusion criteria: No

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1041 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Impact of health mediation on healthcare utilization in people living in informal housing (PLIH) in France | At six months follow-up
  The difference in healthcare utilization by PLIH between groups 2 and group 3
Impact of the intervention on people living in informal housing (PLIH) uptake of organized cancer screening | At six months follow-up
  The difference in organized cancer screening uptake (breast cancer, colorectal cancer, cervical cancer) between PLIH in group 1 and PLIH in group 2
Health mediation conditions required to foster utilization of healthcare services among people living in informal housing (PLIH) in France | At six months follow-up
  The difference in organized cancer screening uptake (at 2 years since diagnosis for breast cancer and colorectal cancer, at 3 years since diagnosis for cervical cancer) between PLIH in group 1 and people living in informal housing in group 3

CONTACTS AND LOCATIONS:
Overall Officials: Judith Martin-Fernandez, PhD, Principal Investigator — Equipe Mérisp/PHARES, INSERM, BPH, U1219, University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No